CLINICAL TRIAL: NCT02581332
Title: The Effects of Mindfulness Meditation on Fibromyalgia-Related Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to insufficient interest in the study and enrollment has been closed
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 32852
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-01

CONDITIONS: Fibromyalgia
Keywords: behavioral intervention
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral: Mindfulness Meditation (Other): Training will be held in groups of up to five participants. All of the participants within this group will receive up to 6 days (20m/d) of meditation training to be administered over 15 days. This is a paradigm similar to one employed in previous studies.
  Interventions: Behavioral: Mindfulness Meditation Training

INTERVENTIONS:
Behavioral: Mindfulness Meditation Training — Training will be held in groups of up to five participants. All of the participants within this group will receive up to 6 days (20m/d) of meditation training to be administered over 15 days. This is a paradigm similar to one employed in previous studies.

SUMMARY:
The purpose of this study is to examine the effects of a brief mindfulness meditation intervention on clinical and experimental pain in fibromyalgia (FM) patients as compared to a wait-list control condition. Based on prior research, investigators' working hypothesis is that this intervention will decrease the severity of FM-associated clinical pain and experimentally induced pain in comparison to pre-intervention scores and a wait-list control group. Additionally, based on prior work, investigators postulate that mindfulness meditation training will decrease a) depression, b) state anxiety, c) overall disease severity, and d) perceived stress, while increasing e) quality of sleep, and f) mindfulness skills in comparison to pre-intervention scores and the wait-list control group.

Investigators will also be testing if decreases in pain ratings during meditation correspond to increases in parasympathetic activity. The relative systemic contributions of the parasympathetic and sympathetic branches of the Autonomic Nervous System (ANS) can be examined by measuring heart rate variability (HRV), or the variability in the beat-to-beat interval. Fast acting, parasympathetically-mediated high frequency (HF) changes in heart rate variability (HF HRV; 0.15-0.40 Hz) provide a reliable indicator of parasympathetic activity. Importantly, decreased HF HRV correlates with increased pain. Investigators therefore will employ psychophysical and physiological methodologies to test the hypothesis that the analgesic effects of mindfulness meditation in FM patients are associated with increases in HF HRV.

DETAILED DESCRIPTION:
Mindfulness and FM-Related Clinical Pain

The lack of clinical improvement in FM patients in response to pharmacologic therapy provides support for the development and validation of cost-effective, narcotic free, cognitive approaches to treating FM.

If the benefits of mindfulness-based interventions can be realized after brief mental training, then this technique could better facilitate treatment in pain patients and become more attractive to clinicians and health insurers. To this extent, investigators have previously shown that four days (20m/d) of mindfulness meditation training in healthy subjects significantly reduced experimental pain unpleasantness by 57% and pain intensity by 40% when compared to rest. Additionally, investigators found that four days of mindfulness-based mental training significantly reduced state anxiety, and these results were realized even after one meditation session. However, it remains unclear if brief mindfulness-based mental training can reliably reduce clinical pain in FM patients. To this extent, investigators will test the efficacy of a brief, mindfulness meditation intervention on FM-related pain. Providing a short, but potentially effective intervention could offset the physical, temporal, and financial barriers to treatment in FM patients.

Mindfulness and FM-Related Experimental Pain

FM patients have been found to have lower pain thresholds across multiple noxious stimulation modalities and suffer from hyperalgesia, an increased sensitivity to pain. While pain thresholds correspond to the point at which a stimulus is experienced as painful, sensitivity to pain refers to an individual's subjective experience of a noxious stimulus. Unfortunately, no known studies have examined the effects of mindfulness meditation on FM-related heat pain thresholds and heat pain sensitivity. The employment of experimentally induced pain manipulations could provide the means to disentangle the constellation of interactions that affect the subjective experience of FM-related pain. To this extent, in addition to examining the effects of mindfulness meditation on clinical pain, investigators will also employ psychophysical methodologies to determine if mindfulness meditation attenuates experimentally induced pain in FM patients.

Heart Rate Variability (HRV) and Fibromyalgia

The Autonomic Nervous System (ANS) is critical for control of homeostatic measures such as blood pressure, body temperature, and heart rate. HRV, or the variability in the beat-to-beat interval, can be used to assess the systemic relative contributions of the parasympathetic and sympathetic branches of the ANS. Parasympathetic effects on heart rate are mediated through the vagus nerve relatively quickly, thus classifying high frequency changes in heart rate (HF HRV; 0.15-0.40 Hz) as a marker of parasympathetic activity.

Interestingly, decreased HF HRV can provide a robust physiological correlate of the subjective experience of pain. In fact, decreased HF HRV is directly associated with a number of clinical pain conditions including fibromyalgia. Additionally, recent findings have shown that meditation directly increases HF HRV. Investigators therefore will employ psychophysical and physiological methodologies to test the hypothesis that the analgesic effects of mindfulness meditation in FM patients are associated with increases in HF HRV.

Specific Aims

To examine the effects of a brief mindfulness meditation intervention on clinical pain (the primary outcome) and experimental pain (the secondary outcome) in FM patients as compared to a wait-list control condition. Investigators will also examine if the analgesic effects of mindfulness meditation are correlated with increases in HF HRV.

Hypotheses

Investigators hypothesize that a brief mindfulness meditation intervention will decrease clinical and experimental pain in FM patients when compared to a wait-list control condition. Investigators hypothesize that the analgesic effects of meditation will be correlated with increases in HF HRV. Investigators also predict that meditation will decrease depression, state anxiety, overall disease severity, and perceived stress, while increasing quality of sleep, and mindfulness skills in comparison to pre-intervention scores and the wait-list control group.

Study Objectives

Primary Objective: The primary objective of this study is to determine if a brief mindfulness meditation intervention can improve FM-related clinical pain. Based on prior research, investigators' working hypothesis is that this intervention will decrease the severity of FM-associated pain in comparison to pre-intervention scores and a wait-list control group.

Secondary Objective: The secondary objective of this study is to determine if a brief mindfulness-based meditation intervention can impact a number of factors associated with FM while proving to be a feasible intervention for this patient population, as measured by an attrition rate of less than 25%. First, investigators will test the hypothesis that mindfulness meditation, in comparison to the wait-list control group and pre-intervention experimental pain ratings, will reduce the subjective experience of experimentally induced pain in FM patients. Specifically, based on preliminary studies, investigators hypothesize that a brief mindfulness meditation intervention will decrease heat pain sensitivity and increase heat pain thresholds in this patient population (see Interventions and Interactions). Additionally, investigators will test the hypothesis that the decreases in clinical and/or experimental pain caused by mindfulness meditation will be associated with increases in HF HRV. Finally, investigators will test if a brief mindfulness-based meditation intervention can improve psychological disposition in FM patients. Based on prior work, investigators postulate that mindfulness meditation training will decrease a) depression, b) state anxiety, c) overall disease severity, and d) perceived stress, while increasing e) quality of sleep, and f) mindfulness skills in comparison to pre-intervention scores and the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Sixty individuals (18-65 years old; male and female) of all ethnic backgrounds will be examined.
* Participants should meet the 2010 revised American College of Rheumatology (ACR) criteria for FM.
* Additionally, only patients who have been on the same medication regimen for FM for the past four weeks will be included.
* Patients must also report a score of greater than or equal to 50 on the Revised FM Impact Questionnaire (FIQR) and a score of less than 20 on the Patient Health Questionnaire-8 (PHQ-8) to be included in the study.
* Importantly, Dr. Dennis Ang will confirm FM diagnoses.

Exclusion Criteria:

* Individuals with chronic heart or lung conditions, who are pregnant, smoke, are currently waiting for a response to an application for disability, have been diagnosed with schizophrenia, bipolar, or any other mental illness or personality disorder, or are planning on undergoing any major elective surgery in the next three months will be excluded.
* Additionally, those patients who have ever meditated (excluding yoga) will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Clinical Pain | 17 days
  Investigators will use "pre-intervention" vs. "post-intervention" VAS overall pain ratings for the previous two weeks (those obtained from sessions 1 and 8, respectively) to test the hypothesis that a mindfulness meditation intervention will decrease clinical pain in FM patients. Investigators will employ a 2 (meditation vs. control) X 2 ("pre" vs. "post-intervention") repeated measures ANOVA (RM ANOVA) to test hypothesized differences between groups. Follow-up post-hocs will be conducted to test significant main effects and interactions.

SECONDARY OUTCOMES:
Experimental Pain | 17 days
  Heat Pain Sensitivity Testing: Investigators will examine data corresponding to the pre and post intervention sessions separately. Investigators will employ a univariate ANOVA to assess if there are baseline differences in pain between groups. With respect to the post-intervention session, investigators will employ a 2 (group) X 2 (rest vs. control/meditation) RM ANOVA to test the hypothesis that meditation will reduce pain ratings when compared to rest and the control group. Follow-up post-hoc tests will be conducted to examine significant main effects and interactions.
  Heat Pain Threshold Testing: In order to test the hypothesis that heat pain thresholds will increase after meditation training and when compared to the wait-list control group, investigators will conduct a 2 (group) X 2 ("pre" vs. "post-intervention") RM ANOVA. Follow-up post-hocs will be conducted to test significant main effects and interactions.
Fibromyalgia-associated symptoms | 17 days
  Investigators will use "pre" vs. "post" ratings (those obtained at sessions 1 and 8, respectively) on the BPI, PHQ-8, CES-D, FIQR, PSS, PCS, PSQI, MASQ, and FMI to test the hypothesis that mindfulness meditation decreases a) pain-related measures, b) depression, c) disease severity d) perceived stress, and e) pain catastrophizing while increasing f) quality of sleep, g) cognitive function, and h) mindfulness ratings. Investigators will use a 2 (group) X 2 ("pre" vs. "post-intervention") RM ANOVA for each of these scales to test the hypotheses. Follow-up post-hocs will be conducted to test significant main effects and interactions.
Fibromyalgia-associated anxiety | 17 days
  In order to test the hypothesis that mindfulness meditation will reduce SAI scores, investigators will perform a 7 (experimental sessions employing meditation) X 2 ("pre" vs. "post") RM ANOVA where "pre" corresponds to SAI scores prior to each intervention and "post" corresponds to SAI scores after each intervention. Follow-up post-hocs will be conducted to test significant main effects and interactions.
High Frequency Heart Rate Variability (HF HRV) | 17 days
  Separate multiple regression models (one for pain intensity and one for pain unpleasantness ratings) will be conducted to test the hypothesis that the analgesic effects of mindfulness meditation will be associated with increases in HF HRV. The regression model(s) will examine if group (wait-list control; meditation) is uniquely associated with the overall model examining the proposed relationship between pain ratings and HF HRV, respectively. Investigators will conduct similar regression models for heat pain thresholds, where the temperature at which a patient first feels pain during session 8 is entered as the dependent variable in the regression model. Investigators will also conduct a similar regression model for clinical pain, where session 8 VAS ratings (intensity and unpleasantness) relating to pain over the previous 2 weeks are entered as the dependent variable, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Fadel Zeidan, PhD, Principal Investigator — Wake Forest University Health Sciences; Dennis Ang, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abeles AM, Pillinger MH, Solitar BM, Abeles M. Narrative review: the pathophysiology of fibromyalgia. Ann Intern Med. 2007 May 15;146(10):726-34. doi: 10.7326/0003-4819-146-10-200705150-00006. PMID 17502633
- [Background] Ang DC, Kaleth AS, Bigatti S, Mazzuca SA, Jensen MP, Hilligoss J, Slaven J, Saha C. Research to encourage exercise for fibromyalgia (REEF): use of motivational interviewing, outcomes from a randomized-controlled trial. Clin J Pain. 2013 Apr;29(4):296-304. doi: 10.1097/AJP.0b013e318254ac76. PMID 23042474
- [Background] Arnold LM, Lu Y, Crofford LJ, Wohlreich M, Detke MJ, Iyengar S, Goldstein DJ. A double-blind, multicenter trial comparing duloxetine with placebo in the treatment of fibromyalgia patients with or without major depressive disorder. Arthritis Rheum. 2004 Sep;50(9):2974-84. doi: 10.1002/art.20485. PMID 15457467
- [Background] Arroyo JF, Cohen ML. Abnormal responses to electrocutaneous stimulation in fibromyalgia. J Rheumatol. 1993 Nov;20(11):1925-31. PMID 7848390
- [Background] Backhaus J, Junghanns K, Broocks A, Riemann D, Hohagen F. Test-retest reliability and validity of the Pittsburgh Sleep Quality Index in primary insomnia. J Psychosom Res. 2002 Sep;53(3):737-40. doi: 10.1016/s0022-3999(02)00330-6. PMID 12217446
- [Background] Bair MJ, Matthias MS, Nyland KA, Huffman MA, Stubbs DL, Kroenke K, Damush TM. Barriers and facilitators to chronic pain self-management: a qualitative study of primary care patients with comorbid musculoskeletal pain and depression. Pain Med. 2009 Oct;10(7):1280-90. doi: 10.1111/j.1526-4637.2009.00707.x. PMID 19818038
- [Background] Bennett RM, Bushmakin AG, Cappelleri JC, Zlateva G, Sadosky AB. Minimal clinically important difference in the fibromyalgia impact questionnaire. J Rheumatol. 2009 Jun;36(6):1304-11. doi: 10.3899/jrheum.081090. Epub 2009 Apr 15. PMID 19369473
- [Background] Black DS, O'Reilly GA, Olmstead R, Breen EC, Irwin MR. Mindfulness meditation and improvement in sleep quality and daytime impairment among older adults with sleep disturbances: a randomized clinical trial. JAMA Intern Med. 2015 Apr;175(4):494-501. doi: 10.1001/jamainternmed.2014.8081. PMID 25686304
- [Background] Buhrman M, Skoglund A, Husell J, Bergstrom K, Gordh T, Hursti T, Bendelin N, Furmark T, Andersson G. Guided internet-delivered acceptance and commitment therapy for chronic pain patients: a randomized controlled trial. Behav Res Ther. 2013 Jun;51(6):307-15. doi: 10.1016/j.brat.2013.02.010. Epub 2013 Mar 14. PMID 23548250
- [Background] Chaves JF, Brown JM. Spontaneous cognitive strategies for the control of clinical pain and stress. J Behav Med. 1987 Jun;10(3):263-76. doi: 10.1007/BF00846540. PMID 3612783
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] Coghill RC, Eisenach J. Individual differences in pain sensitivity: implications for treatment decisions. Anesthesiology. 2003 Jun;98(6):1312-4. doi: 10.1097/00000542-200306000-00003. No abstract available. PMID 12766637
- [Background] Coghill RC, McHaffie JG, Yen YF. Neural correlates of interindividual differences in the subjective experience of pain. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8538-42. doi: 10.1073/pnas.1430684100. Epub 2003 Jun 24. PMID 12824463
- [Background] Cohen BH, Lea RB (2004) Essentials of statistics for the social and behavioral sciences. Hoboken, N.J.: Wiley.
- [Background] Cohen S, Williamson, G. (1988) Perceived stress in a probability sample of the United States. Newbury Park, CA: Sage.
- [Background] Cuijpers P, van Straten A, Andersson G. Internet-administered cognitive behavior therapy for health problems: a systematic review. J Behav Med. 2008 Apr;31(2):169-77. doi: 10.1007/s10865-007-9144-1. PMID 18165893
- [Background] Davis MC, Zautra AJ. An online mindfulness intervention targeting socioemotional regulation in fibromyalgia: results of a randomized controlled trial. Ann Behav Med. 2013 Dec;46(3):273-84. doi: 10.1007/s12160-013-9513-7. PMID 23670111
- [Background] Eccleston C, Fisher E, Craig L, Duggan GB, Rosser BA, Keogh E. Psychological therapies (Internet-delivered) for the management of chronic pain in adults. Cochrane Database Syst Rev. 2014 Feb 26;2014(2):CD010152. doi: 10.1002/14651858.CD010152.pub2. PMID 24574082
- [Background] Ferrari R, Russell AS. A questionnaire using the modified 2010 American College of Rheumatology criteria for fibromyalgia: specificity and sensitivity in clinical practice. J Rheumatol. 2013 Sep;40(9):1590-5. doi: 10.3899/jrheum.130367. Epub 2013 Jul 1. PMID 23818707
- [Background] Fjorback LO, Arendt M, Ornbol E, Walach H, Rehfeld E, Schroder A, Fink P. Mindfulness therapy for somatization disorder and functional somatic syndromes: randomized trial with one-year follow-up. J Psychosom Res. 2013 Jan;74(1):31-40. doi: 10.1016/j.jpsychores.2012.09.006. Epub 2012 Oct 1. PMID 23272986
- [Background] Gardner-Nix J, Backman S, Barbati J, Grummitt J. Evaluating distance education of a mindfulness-based meditation programme for chronic pain management. J Telemed Telecare. 2008;14(2):88-92. doi: 10.1258/jtt.2007.070811. PMID 18348755
- [Background] Gibson SJ, Littlejohn GO, Gorman MM, Helme RD, Granges G. Altered heat pain thresholds and cerebral event-related potentials following painful CO2 laser stimulation in subjects with fibromyalgia syndrome. Pain. 1994 Aug;58(2):185-193. doi: 10.1016/0304-3959(94)90198-8. PMID 7816486
- [Background] Giesecke T, Gracely RH, Williams DA, Geisser ME, Petzke FW, Clauw DJ. The relationship between depression, clinical pain, and experimental pain in a chronic pain cohort. Arthritis Rheum. 2005 May;52(5):1577-84. doi: 10.1002/art.21008. PMID 15880832
- [Background] Griffiths F, Lindenmeyer A, Powell J, Lowe P, Thorogood M. Why are health care interventions delivered over the internet? A systematic review of the published literature. J Med Internet Res. 2006 Jun 23;8(2):e10. doi: 10.2196/jmir.8.2.e10. PMID 16867965
- [Background] Grossman P, Tiefenthaler-Gilmer U, Raysz A, Kesper U. Mindfulness training as an intervention for fibromyalgia: evidence of postintervention and 3-year follow-up benefits in well-being. Psychother Psychosom. 2007;76(4):226-33. doi: 10.1159/000101501. PMID 17570961
- [Background] Hays B (2008) A practical security analysis. In: SANS Institute.
- [Background] Hurtig IM, Raak RI, Kendall SA, Gerdle B, Wahren LK. Quantitative sensory testing in fibromyalgia patients and in healthy subjects: identification of subgroups. Clin J Pain. 2001 Dec;17(4):316-22. doi: 10.1097/00002508-200112000-00005. PMID 11783811
- [Background] Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK91497/ PMID 22553896
- [Background] Julien N, Goffaux P, Arsenault P, Marchand S. Widespread pain in fibromyalgia is related to a deficit of endogenous pain inhibition. Pain. 2005 Mar;114(1-2):295-302. doi: 10.1016/j.pain.2004.12.032. PMID 15733656
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn J (1990) Full Catastrophe Living. New York: Delta Trade Paperbacks.
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Kosek E, Ekholm J, Hansson P. Modulation of pressure pain thresholds during and following isometric contraction in patients with fibromyalgia and in healthy controls. Pain. 1996 Mar;64(3):415-423. doi: 10.1016/0304-3959(95)00112-3. PMID 8783304
- [Background] Koyama T, McHaffie JG, Laurienti PJ, Coghill RC. The subjective experience of pain: where expectations become reality. Proc Natl Acad Sci U S A. 2005 Sep 6;102(36):12950-5. doi: 10.1073/pnas.0408576102. Epub 2005 Sep 6. PMID 16150703
- [Background] Kozasa EH, Tanaka LH, Monson C, Little S, Leao FC, Peres MP. The effects of meditation-based interventions on the treatment of fibromyalgia. Curr Pain Headache Rep. 2012 Oct;16(5):383-7. doi: 10.1007/s11916-012-0285-8. PMID 22717699
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Lauche R, Cramer H, Dobos G, Langhorst J, Schmidt S. A systematic review and meta-analysis of mindfulness-based stress reduction for the fibromyalgia syndrome. J Psychosom Res. 2013 Dec;75(6):500-10. doi: 10.1016/j.jpsychores.2013.10.010. Epub 2013 Oct 26. PMID 24290038
- [Background] Lobanov OV, Quevedo AS, Hadsel MS, Kraft RA, Coghill RC. Frontoparietal mechanisms supporting attention to location and intensity of painful stimuli. Pain. 2013 Sep;154(9):1758-1768. doi: 10.1016/j.pain.2013.05.030. Epub 2013 May 24. PMID 23711484
- [Background] Lobanov OV, Zeidan F, McHaffie JG, Kraft RA, Coghill RC. From cue to meaning: brain mechanisms supporting the construction of expectations of pain. Pain. 2014 Jan;155(1):129-136. doi: 10.1016/j.pain.2013.09.014. Epub 2013 Sep 17. PMID 24055334
- [Background] Moore A, Malinowski P. Meditation, mindfulness and cognitive flexibility. Conscious Cogn. 2009 Mar;18(1):176-86. doi: 10.1016/j.concog.2008.12.008. Epub 2009 Jan 31. PMID 19181542
- [Background] Morone NE, Greco CM, Weiner DK. Mindfulness meditation for the treatment of chronic low back pain in older adults: a randomized controlled pilot study. Pain. 2008 Feb;134(3):310-319. doi: 10.1016/j.pain.2007.04.038. Epub 2007 Jun 1. PMID 17544212
- [Background] Murray E, Burns J, See TS, Lai R, Nazareth I. Interactive Health Communication Applications for people with chronic disease. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD004274. doi: 10.1002/14651858.CD004274.pub4. PMID 16235356
- [Background] Oshiro Y, Quevedo AS, McHaffie JG, Kraft RA, Coghill RC. Brain mechanisms supporting spatial discrimination of pain. J Neurosci. 2007 Mar 28;27(13):3388-94. doi: 10.1523/JNEUROSCI.5128-06.2007. PMID 17392455
- [Background] Price DD. Psychological and neural mechanisms of the affective dimension of pain. Science. 2000 Jun 9;288(5472):1769-72. doi: 10.1126/science.288.5472.1769. PMID 10846154
- [Background] Price DD, McHaffie JG, Larson MA. Spatial summation of heat-induced pain: influence of stimulus area and spatial separation of stimuli on perceived pain sensation intensity and unpleasantness. J Neurophysiol. 1989 Dec;62(6):1270-9. doi: 10.1152/jn.1989.62.6.1270. PMID 2600624
- [Background] Radloff LS (1977) The CES-D scale: a self-report depression scale for research in the general population. Applied Psychological Measurement 1.
- [Background] Rosier EM, Iadarola MJ, Coghill RC. Reproducibility of pain measurement and pain perception. Pain. 2002 Jul;98(1-2):205-16. doi: 10.1016/s0304-3959(02)00048-9. PMID 12098633
- [Background] Schmidt S, Grossman P, Schwarzer B, Jena S, Naumann J, Walach H. Treating fibromyalgia with mindfulness-based stress reduction: results from a 3-armed randomized controlled trial. Pain. 2011 Feb;152(2):361-369. doi: 10.1016/j.pain.2010.10.043. Epub 2010 Dec 13. PMID 21146930
- [Background] Seidenberg M, Haltiner A, Taylor MA, Hermann BB, Wyler A. Development and validation of a Multiple Ability Self-Report Questionnaire. J Clin Exp Neuropsychol. 1994 Feb;16(1):93-104. doi: 10.1080/01688639408402620. PMID 8150893
- [Background] Sephton SE, Salmon P, Weissbecker I, Ulmer C, Floyd A, Hoover K, Studts JL. Mindfulness meditation alleviates depressive symptoms in women with fibromyalgia: results of a randomized clinical trial. Arthritis Rheum. 2007 Feb 15;57(1):77-85. doi: 10.1002/art.22478. PMID 17266067
- [Background] Skaer TL. Fibromyalgia: disease synopsis, medication cost effectiveness and economic burden. Pharmacoeconomics. 2014 May;32(5):457-66. doi: 10.1007/s40273-014-0137-y. PMID 24504852
- [Background] Spielberger CD, Goruch, R.L., Lushene, R., Vagg, P.R. Jacobs, G.A. (1983) Manual for the state-trati anxiety inventory. Palo Alt, CA: Consulting Psychologists Press.
- [Background] Starr CJ, Sawaki L, Wittenberg GF, Burdette JH, Oshiro Y, Quevedo AS, Coghill RC. Roles of the insular cortex in the modulation of pain: insights from brain lesions. J Neurosci. 2009 Mar 4;29(9):2684-94. doi: 10.1523/JNEUROSCI.5173-08.2009. PMID 19261863
- [Background] Sullivan MJL, Bishop SR, Pivik J (1995) The Pain Catastrophizing Scale: Development and validation. Psychol Assessment 7:524-532.
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Turk DC, Robinson JP, Burwinkle T. Prevalence of fear of pain and activity in patients with fibromyalgia syndrome. J Pain. 2004 Nov;5(9):483-90. doi: 10.1016/j.jpain.2004.08.002. PMID 15556826
- [Background] Walach H, Buchheld N, Buttenmuller V, Kleinknecht N, Schmidt S (2006) Measuring mindfulness - the Freiburg Mindfulness Inventory (FMI). Pers Indiv Differ 40:1543-1555.
- [Background] Walitt B, Fitzcharles MA, Hassett AL, Katz RS, Hauser W, Wolfe F. The longitudinal outcome of fibromyalgia: a study of 1555 patients. J Rheumatol. 2011 Oct;38(10):2238-46. doi: 10.3899/jrheum.110026. Epub 2011 Jul 15. PMID 21765102
- [Background] Williams DA, Arnold LM. Measures of fibromyalgia: Fibromyalgia Impact Questionnaire (FIQ), Brief Pain Inventory (BPI), Multidimensional Fatigue Inventory (MFI-20), Medical Outcomes Study (MOS) Sleep Scale, and Multiple Ability Self-Report Questionnaire (MASQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S86-97. doi: 10.1002/acr.20531. No abstract available. PMID 22588773
- [Background] Wolfe F, Brahler E, Hinz A, Hauser W. Fibromyalgia prevalence, somatic symptom reporting, and the dimensionality of polysymptomatic distress: results from a survey of the general population. Arthritis Care Res (Hoboken). 2013 May;65(5):777-85. doi: 10.1002/acr.21931. PMID 23424058
- [Background] Yarnitsky D, Sprecher E. Thermal testing: normative data and repeatability for various test algorithms. J Neurol Sci. 1994 Aug;125(1):39-45. doi: 10.1016/0022-510x(94)90239-9. PMID 7964887
- [Background] Yelle MD, Oshiro Y, Kraft RA, Coghill RC. Temporal filtering of nociceptive information by dynamic activation of endogenous pain modulatory systems. J Neurosci. 2009 Aug 19;29(33):10264-71. doi: 10.1523/JNEUROSCI.4648-08.2009. PMID 19692600
- [Background] Zeidan F, Gordon NS, Merchant J, Goolkasian P. The effects of brief mindfulness meditation training on experimentally induced pain. J Pain. 2010 Mar;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015. Epub 2009 Oct 22. PMID 19853530
- [Background] Zeidan F, Johnson SK, Gordon NS, Goolkasian P. Effects of brief and sham mindfulness meditation on mood and cardiovascular variables. J Altern Complement Med. 2010 Aug;16(8):867-73. doi: 10.1089/acm.2009.0321. PMID 20666590
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Zeidan F, Martucci KT, Kraft RA, McHaffie JG, Coghill RC. Neural correlates of mindfulness meditation-related anxiety relief. Soc Cogn Affect Neurosci. 2014 Jun;9(6):751-9. doi: 10.1093/scan/nst041. Epub 2013 Apr 24. PMID 23615765
- [Background] Zeidan F, Martucci KT, Kraft RA, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. J Neurosci. 2011 Apr 6;31(14):5540-8. doi: 10.1523/JNEUROSCI.5791-10.2011. PMID 21471390